CLINICAL TRIAL: NCT06829641
Title: A Multicenter Real-World Data Pooled Analysis: The Clinical Outcomes of Tislelizumab Combined With Chemotherapy as Induction Therapy in Stage III (cTNM-IIIB/IIIC) NSCLC
Brief Title: Clinical Outcomes of Tislelizumab Combined With Chemotherapy as Induction Therapy in Stage III (cTNM-IIIB/IIIC) NSCLC
Status: Not yet recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhou Qinghua, Academic Director of the Lung Cancer Center at West China Hospital, Sichuan Universit, West China Hospital
Other Study IDs: CLOG-0004
Record Dates: First submitted 2025-02-09; First posted 2025-02-17 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: NSCLC Stage IIIB, NSCLC Stage IIIC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Tislelizumab Combined with Chemotherapy, — Tislelizumab Combined with Chemotherapy as Induction Therapy

SUMMARY:
This is an observational study evaluating the clinical characteristics, treatment patterns, and clinical outcomes in Stage III (cTNM-IIIB/IIIC) Non-Small Cell Lung Cancer.Patients meeting inclusion and exclusion criteria were enrolled, with treatment modalities and clinical outcomes of stage III non-small cell lung cancer (NSCLC) patients from multiple tertiary hospitals in real-world settings since August 2020 being collected and analyzed.

DETAILED DESCRIPTION:
Key Inclusion Population： Stage IIIB/IIIC NSCLC patients confirmed by histological or cytological examination based on the 8th edition of the AJCC staging system.Patients were negative for EGFR-sensitive mutations or ALK/ROS1 fusion alterations.

No prior chemotherapy, radiotherapy, surgical intervention, or immunotherapy had been administered.ECOG PS scores of the enrolled patients ranged from 0 to 2.

Neoadjuvant/Induction Therapy Regimen:

Tislelizumab combined with platinum-based doublet chemotherapy was administered for at Least Two Cycles , followed by surgical resection or other therapeutic interventions (e.g., radiotherapy/chemotherapy). Real-world clinical outcomes were collected and analyzed based on patients' subsequent treatment pathways.Clinical Stage IIIB-IIIC Non-Small Cell Lung Cancer (AJCC 8th Edition Staging); ECOG PS Score 0-2

Retrospective data collection was conducted for cases prior to site initiation, while prospective collection was implemented for post-initiation cases.

Collected parameters include:

1. Patient clinical characteristics
2. Treatment patterns
3. Treatment compliance
4. Safety profiles
5. Event-free survival (EFS) and overall survival (OS) tracking

ELIGIBILITY:
Inclusion Criteria:

Stage IIIB/IIIC NSCLC patients confirmed by histological or cytological examination based on the 8th edition of the AJCC staging system.

Patients were negative for EGFR-sensitive mutations or ALK/ROS1 fusion alterations.

No prior chemotherapy, radiotherapy, surgical intervention, or immunotherapy had been administered.

ECOG PS scores of the enrolled patients ranged from 0 to 2.

Exclusion Criteria:

Patients with other previous malignancies did not require additional treatment. Patients with incomplete key baseline and treatment information:including clinical stage, pathological type, neoadjuvant treatment, pathological response, imaging response after neoadjuvant.

Patients included in anti-tumor drug intervention or unblinded clinical trials, in which the treatment being administered is unknown.

Prior surgery, radiotherapy or systemic therapy for NSCLC, including radiofrequency ablation, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stage IIIB/IIIC NSCLC patients confirmed by histological or cytological examination based on the 8th edition of the AJCC staging system.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-09 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
major pathological response | ;usually 1 week after surgery
  viable tumor cell less than 10%

SECONDARY OUTCOMES:
R0 resection rate | ,usually 1 week after surgery
  margin negative resection
Down-staging rate | usually 1 week after surgery
  clinical and pathological downstaging
Impact of Neoadjuvant Therapy on Surgical Outcomes | usually 1 week after surgery
  Surgical Rate
The outcome of survival | usually 12 month after Induction Therapy
  patterns and Outcomes of Postoperative Disease Recurrence/Progression
12month event-free survival rate | rom date of diagnosis until the date of first documented progression, the rate of recurrence or date of death from any cause, whichever came first, assessed up to 12 months
  the time from randomization to any progression of disease precluding surgery, progresson or recurrence of disease after surgery, progression of disease in the absence of surgery, or death from any cases;
OS | from date of diagnosis until the date of death from any cause, whichever came first, assessed up to 60 months
  From diagnosis to the death;

IPD SHARING:
Plan to Share IPD: No